CLINICAL TRIAL: NCT00007813
Title: TREATMENT OF CHILDREN AND YOUNG ADULTS WITH RECURRENT/REFRACTORY SOLID TUMORS WITH HIGH DOSE ETOPOSIDE AND CARBOPLATIN PLUS ESCALATING DOSE CYCLOPHOSPHAMIDE, FOLLOWED BY HEMATOPOIETIC RESCUE USING AUTOLOGOUS CD34+ SELECTED BLOOD STEM CELLS: A PILOT STUDY
Brief Title: Peripheral Stem Cell Transplantation Plus Chemotherapy in Treating Patients With Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Amgen (Industry); Baxter Healthcare Corporation (Industry); Nexell Therapeutics Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JHOC-9512; CDR0000064263 (Registry Identifier: PDQ (Physician Data Query)); NCI-V95-0688 (Registry Identifier: other); 94-12-23-02 (Other: JHM IRB)
Record Dates: First submitted 2001-01-06; First posted 2004-04-02 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Liver Cancer; Neuroblastoma; Ovarian Cancer; Sarcoma; Testicular Germ Cell Tumor
Keywords: recurrent childhood rhabdomyosarcoma; childhood craniopharyngioma; recurrent childhood brain tumor; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; stage IV childhood liver cancer; recurrent childhood liver cancer; childhood hepatoblastoma; childhood central nervous system germ cell tumor; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; childhood germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; extragonadal germ cell tumor; childhood oligodendroglioma; childhood choroid plexus tumor; childhood grade III meningioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; previously treated childhood rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood ependymoma; childhood teratoma; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood extragonadal germ cell tumor; recurrent childhood malignant germ cell tumor; childhood atypical teratoid/rhabdoid tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Liver Neoplasms; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Testicular Germ Cell Tumor; Hepatoblastoma; Testicular Neoplasms; Oligodendroglioma; Choroid Plexus Neoplasms; Astrocytoma; Medulloblastoma; Optic Nerve Glioma; Neuroectodermal Tumors, Primitive, Peripheral; Familial ependymoma; Teratoma; Ovarian Germ Cell Cancer; Rhabdoid Tumor | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cyclophosphamide; Drug: etoposide; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of cyclophosphamide when given together with combination chemotherapy and a peripheral stem cell transplant in treating patients with malignant solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether autologous transplantation of mobilized CD34+ peripheral blood stem cells (PBSC) can provide complete hematologic reconstitution after myeloablative chemotherapy comprising etoposide (VP-16) and carboplatin (CBDCA) in patients with metastatic or recurrent rhabdomyosarcoma, neuroblastoma, Ewing's sarcoma/primitive neuroectodermal tumor, germ cell tumors, childhood brain tumors, or hepatoblastoma.
* Determine the frequency and yield of CD34+ PBSC and granulocyte-macrophage colony-forming units (GM-CFU) that are mobilized, harvested, and purified after a single priming course of high-dose cyclophosphamide (CTX) followed by filgrastim (G-CSF).
* Correlate the number of CD34+ cells and GM-CFU in the autologous PBSC graft with time to engraftment of white blood cells, neutrophils, and platelets in these patients.
* Determine the optimal day of PBSC harvest after a single priming course of high-dose CTX and G-CSF in these patients.
* Determine whether CD34+ PBSC rescue and daily post-transplantation G-CSF decrease the time to hematopoietic recovery after high-dose VP-16 and CBDCA compared to historical results achieved in similar patients rescued with bone marrow.
* Compare the tumor cell content of marrow, mobilized blood, and purified CD34+ PBSC graft preparations.
* Determine the optimal timing of PBSC mobilization and harvest in relation to extent of prior chemotherapy in these patients.
* Determine the feasibility of a single leukapheresis for PBSC harvest in children.
* Determine the toxic effects of this regimen in these patients.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of cyclophosphamide.

Mobilization/harvest: Patients receive cyclophosphamide IV over 90 minutes on day 0 and filgrastim (G-CSF) subcutaneously or IV over 30 minutes on days 2-15 or until blood counts recover. Peripheral blood stem cells (PBSC) are harvested and selected for CD34+ cells on day 15. Bone marrow is also harvested in case insufficient PBSC are harvested.

Preparative regimen/transplantation: Patients receive carboplatin IV over 1 hour and etoposide IV continuously on days -6 to -4. Cyclophosphamide is administered IV over 1 hour on days -3 and -2 or IV continuously on days -3 and -2, -4 to -2, -5 to -2, or -6 to -2. PBSC or bone marrow is reinfused on day 0.

Cohorts of 3-10 patients receive escalating doses of cyclophosphamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the highest dose at which 20% of patients experience dose-limiting toxicity.

At least 6 additional patients receive cyclophosphamide at the MTD.

PROJECTED ACCRUAL: A minimum of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignant solid tumor, including any of the following:

  * Rhabdomyosarcoma
  * Neuroblastoma
  * Ewing's sarcoma/primitive neuroectodermal tumor
  * Germ cell tumors
  * Childhood brain tumors
  * Hepatoblastoma
* Metastatic disease OR has failed at least first-line therapy
* Ineligible for higher priority protocols

PATIENT CHARACTERISTICS:

Age:

* Under 36 at transplantation

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 75,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Liver function tests no greater than 2 times normal OR
* No active hepatitis on liver biopsy
* No hepatitis B infection

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Glomerular filtration rate (preferably measured) greater than 60% of normal

Cardiovascular:

* Left ventricular ejection fraction at least 45%
* No active congestive heart failure
* No active arrhythmia

Pulmonary:

* Age 8 and under: clinically normal pulmonary function
* Over age 8: FEV1 and FVC at least 50% predicted
* Arterial blood gases normal and DLCO at least 50% if spirograms difficult to
* interpret due to poor patient effort, recent surgery, or pulmonary tumor
* involvement

Other:

* No mucositis or mucosal infection prior to myeloablative chemotherapy
* HIV negative
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 1997-05-31 (Actual); Primary Completion 2005-02-01 (Actual); Study Completion 2005-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen R. Chen, MD, PhD, MHS, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Leung W, Chen AR, Klann RC, et al.: Tumor cells frequently detected in marrow and mobilized blood hematopoietic grafts in neuroblastoma and primitive neuroblastoma and primitive neuroectodermal tumor: purging by immunomagnetic CD34+ cell selection. [Abstract] Blood 88: A-1917, 482a, 1996.
- [Background] Chen AR, Cohen KJ, Eby LL, et al.: Heterogenous mobilization of CD34+ blood stem cells for autologous rescue of children with poor prognosis solid tumors. [Abstract] Blood 86: 403a, 1995.
- [Result] Chen AR, Wiangon S, Noga SJ, et al.: Rapid engraftment of CD34+ selected peripheral blood stem cells (PBSC) after high-dose chemotherapy for patients with recurrent, refractory, or metastatic pediatric solid tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A2038, 530a, 1998.
- [Result] Leung W, Chen AR, Klann RC, Moss TJ, Davis JM, Noga SJ, Cohen KJ, Friedman AD, Small D, Schwartz CL, Borowitz MJ, Wharam MD, Paidas CN, Long CA, Karandish S, McMannis JD, Kastan MB, Civin CI. Frequent detection of tumor cells in hematopoietic grafts in neuroblastoma and Ewing's sarcoma. Bone Marrow Transplant. 1998 Nov;22(10):971-9. doi: 10.1038/sj.bmt.1701471. PMID 9849694